CLINICAL TRIAL: NCT02610231
Title: A Phase 3, Long-term, Open-label Study of Istradefylline in Subjects With Moderate to Severe Parkinson's Disease
Brief Title: Long Term Study of Istradefylline in Subjects With Moderate to Severe Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6002-018
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Moderate to Severe Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Istradefylline 20 mg or 40 mg (Experimental): Treatment for 52 weeks
  Interventions: Drug: Istradefylline 20 mg or 40 mg

INTERVENTIONS:
Drug: Istradefylline 20 mg or 40 mg — Istradefylline 20 or 40 mg
  Other Names: KW-6002

SUMMARY:
This is a Phase 3, 52-week, open-label, flexible-dose, multinational, multicenter study to evaluate the safety and tolerability of istradefylline 20 or 40 mg/d in subjects with moderate to severe PD with motor fluctuations and dyskinesia on levodopa combination (levodopa/carbidopa or levodopa/benserazide) therapy plus at least one adjunctive PD medication. Subjects who completed 12 weeks of double-blind treatment and the 30-day follow-up period in Study No. 6002-014 will undergo Screening and Baseline evaluations for eligibility for the study. Eligible subjects will be treated with istradefylline at a starting dose of 20 mg/d with an option for a dose adjustment to 40 mg/d at Week 12 based on the Investigator's judgment of each subject's response and tolerability. If deemed necessary, one unscheduled dose adjustment visit between Week 2 to Week 12 is allowed in accordance with clinical judgment of the Investigator. Subjects who had a dose adjustment to 40 mg/d can have their dose decreased to 20 mg/d by the Investigator at a second unscheduled dose adjustment visit if there are tolerability issues. The istradefylline dose should remain fixed between Week 26 to Week 52. Consultation with the Sponsor's Medical Monitor is required prior to any unscheduled dose adjustment visits. A subject may discontinue from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Subjects who completed Study No. 6002-014 inclusive of the 30-day follow-up period;
3. Currently taking levodopa combination (carbidopa/levodopa or benserazide/levodopa) therapy plus at least one adjunctive PD medication;
4. Women of child-bearing potential (WOCBP) must use a reliable method of contraception and have a negative serum pregnancy test at Screening;

Exclusion Criteria:

1. Subjects with less than 70% treatment compliance throughout their enrollment on Study No 6002-014 and or with major protocol deviations in Study No. 6002-014 (subjects who failed to meet any of the inclusion criteria, subjects who met any of the exclusion criteria or subjects who met the criteria for subject withdrawal but who were not withdrawn);
2. Subjects on apomorphine and/or dopamine receptor antagonists or direct gastrointestinal levodopa infusion;
3. Subject who have had neurosurgical operation for PD;
4. Subjects taking A2a antagonist, potent CYP3A4 inhibitors, potent CYP34A inducers;
5. Subjects who have had a diagnosis of cancer or evidence of continued malignancy within the past three years (with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ prostate cancer with normal prostate-specific antigens post resection).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyowa Hakko Kirin Pharma, Inc., Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (53):
- United States (23):
  - Kyowa PD Site, Phoenix, Arizona
  - Kyowa PD Site, Sun City, Arizona
  - Kyowa PD Site, Tucson, Arizona
  - Kyowa PD Site, Fountain Valley, California
  - Kyowa PD Site, Los Angeles, California
  - Kyowa PD Site, Oxnard, California
  - Kyowa PD Site, Torrance, California
  - Kyowa PD Site, Englewood, Colorado
  - Kyowa PD Site, Danbury, Connecticut
  - Kyowa PD Site, Boca Raton, Florida
  - Kyowa PD Site, Port Charlotte, Florida
  - Kyowa PD Site, Tampa, Florida
  - Kyowa PD Site, Atlanta, Georgia
  - Kyowa PD Site, Augusta, Georgia
  - Kyowa PD Site, Des Moines, Iowa
  - Kyowa PD Site, Kansas City, Kansas
  - Kyowa PD Site, Boston, Massachusetts
  - Kyowa PD Site, West Bloomfield, Michigan
  - Kyowa PD Site, Albany, New York
  - Kyowa PD Site, New York, New York
  - Kyowa PD Site, Asheville, North Carolina
  - Kyowa PD Site, Durham, North Carolina
  - Kyowa PD Site, Toledo, Ohio
- Canada (2):
  - Kyowa PD Site, Calgary, Alberta
  - Kyowa PD Site, Toronto, Ontario
- Czechia (3):
  - Kwoya PD Site, Brno
  - Kyowa PD Site, Litomyšl
  - Kyowa PD Site, Prague
- Germany (6):
  - Kyowa PD Site, Beelitz-Heilstätten
  - Kyowa PD Site, Bremerhaven
  - Kyowa PD Site, Dresden
  - Kyowa PD Site, Haag
  - Kyowa PD Site, Kassel
  - Kyowa PD Site, München
- Israel (4):
  - Kyowa PD Site, Haifa
  - Kyowa PD Site, Jerusalem
  - Kyowa PD Site, Ramat Gan
  - Kyowa PD Site, Tel Aviv
- Italy (7):
  - Kyowa PD Site, Grosseto
  - Kyowa PD Site, Pavia
  - Kyowa PD Site, Pisa
  - Kyowa PD Site, Roma
  - Kyowa PD Site, Rome
  - Kyowa PD Site, Venezia
  - Kyowa PD Site, Vicenza
- Poland (5):
  - Kyowa PD Site, Bydgoszcz
  - Kyowa PD Site, Krakow
  - Kyowa PD Site, Lublin
  - Kyowa PD Site, Poznan
  - Kyowa PD Site, Warsaw
- Serbia (3):
  - Kyowa PD Site 1, Belgrade
  - Kyowa PD Site 4, Belgrade
  - Kyowa PD Site, Novi Sad

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects must have completed 12 weeks of double blind treatment in study 6002-014 including a 30 day follow up period. All subjects were screened for eligibility to participate in the trial. Subjects that met all the inclusion and none of the exclusion criteria were eligible for entry into the trial.
Groups:
- Istradefylline 20 mg or 40mg: Eligible subjects were treated with istradefylline at a starting dose of 20mg/d with an option for dose adjustment at week 40mg/d at week 12 based on the Investigator's judgement of each subject's response and tolerability. If deemed necessary, one unscheduled dose adjustment visit between weeks 2 and 12 was allowed in accordance with the Investigator's clinical judgement. Subjects who had a dose adjustment to 40 mg/d could have their dose decreased to 20mg/d by the investigator at a second unscheduled dose adjustment visit if there were tolerability issues. The istradefylline dose was to remain fixed between Weeks 26 and weeks 52. Subjects took one tablet orally in the morning
Period: Overall Study
Arm/Group | Istradefylline 20 mg or 40mg
Started | 239
Completed | 179
Not Completed | 60
Not completed — Withdrawal by Subject | 27
Not completed — Adverse Event | 20
Not completed — Death | 5
Not completed — Surgery | 2
Not completed — Physician Decision | 1
Not completed — Non Compliance | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: The study was a 52 week open-label, phase 3 continuation of study 6002-014. Subjects must have completed 12 weeks of double blind treatment including a 30 day follow up period on 6002-014 prior to enrollment in 6002-018.
Groups:
- Istradefylline 20 mg or 40 mg: Treatment for 52 weeks
  Istradefylline 20 mg or 40 mg
Arm/Group | Istradefylline 20 mg or 40 mg
Number analyzed (Participants) | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 123
  >=65 years | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 233
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 6
  United States | 79
  Czechia | 41
  Poland | 49
  Italy | 18
  Israel | 16
  Serbia | 18
  Germany | 12

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Long-term Safety and Tolerability of Oral Istradefylline (20mg or 40mg/Day [mg/d])
Description: The number of subjects experiencing an adverse event as well as clinical laboratory tests (chemistry, haematology and urinalysis) were collected to evaluate the safety profile of istradefylline (20mg or 40mg/day [mg/d]).
Time Frame: From screening through to study completion, an average of 52 weeks
Population: All participants who received at least one dose of assigned study drug (even a partial dose) made up the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Analysis Set: Open label treatment for 52 weeks with Istradefylline 20 mg or 40 mg
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 239
Participants
  Number of participants with any TEAE | 141
  Number of participants who did'nt have any TEAE | 98

2. Secondary Outcome: Patient Global Impression - Overall Condition (Improvement by Study Visit) (ITT Analysis Set).
Description: The number and percentage of subjects showing improvement (moderate or mild) on PGI-I scores with Istradefylline 20 mg or 40 mg. Each subjects 'key symptom' (the symptom they had most trouble with) on the PGI-I was identified and evaluated at baseline and at Week 12, 26 and 52. In addition, the subject's overall condition and symptoms of fatigue, sleep and motivation to get things done were also evaluated at week 12, 26 and 52. Subjects rated each on a scale 1 to 5 for change from baseline status utilizing the following scale: 1= Moderate improvement (or greater) 2= Mild improvement, 3= No change from baseline, 4 = Mild deterioration, 5= Moderate deterioration (or greater).
Time Frame: From baseline through to study completion at week 52, plus 30 days post last dose
Measure: Count of Participants; unit: Participants
Groups:
- Efficacy Analysis Based on PGI-I Scores at Week 12.: The percentage of subjects showing improvement (moderate or mild) on PGI-I scores at (week 12).
- Efficacy Analysis Based on PGI-I Scores at Week 26.: The percentage of subjects showing improvement (moderate or mild) on PGI-I scores at (week 26).
- Efficacy Analysis Based on PGI-I Scores at Week 52.: The percentage of subjects showing improvement (moderate or mild) on PGI-I scores at (week 52).
Arm/Group | Efficacy Analysis Based on PGI-I Scores at Week 12. | Efficacy Analysis Based on PGI-I Scores at Week 26. | Efficacy Analysis Based on PGI-I Scores at Week 52.
Number analyzed (Participants) | 237 | 214 | 187
Participants
  Overall Condition | 115 | 109 | 76
  Fatigue | 68 | 62 | 40
  Sleep | 48 | 61 | 37
  Motivation to get things done | 64 | 66 | 45
  Key Symtom | 97 | 95 | 73

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored and collected for up to 52 weeks from the time subjects signed the ICF and for 30 days after their last dose of study drug.
Arm/Group | Istradefylline 20 mg or 40 mg
All-Cause Mortality (participants affected / at risk) | 5/239
Serious Adverse Events (participants affected / at risk) | 30/239
Other Adverse Events (participants affected / at risk) | 91/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Istradefylline 20 mg or 40 mg (N=239)
Circulatory Collapse (Vascular disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Asthenia (General disorders) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 1 (1)
Procedure Pain (Injury, poisoning and procedural complications) | 2 (2)
Pubis Fracture (Injury, poisoning and procedural complications) | 2 (2)
Incorrect dose Administered (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Protein Total Decrease (Investigations) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
On and Off Phenomenon (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Parkinson's Disease (Nervous system disorders) | 3 (3)
Convulsion (Nervous system disorders) | 1 (1)
Transcient Ischaemic attack (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1)
Multiple Sclerosis (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (2)
Dyskinesia (Nervous system disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Gas Gangrene (Infections and infestations) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Istradefylline 20 mg or 40 mg (N=239)
Dyskinesia (Nervous system disorders) | 43
Fall (Nervous system disorders) | 29
Parkinson's disease (Nervous system disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT02610231/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02610231/SAP_001.pdf